CLINICAL TRIAL: NCT01722656
Title: Open Label Study: Intravitreal Aflibercept Injection for the Treatment of Submacular Vascularized Pigment Epithelial Detachment.
Brief Title: Intravitreal Aflibercept Injection for the Treatment of Submacular Vascularized Pigment Epithelial Detachment
Acronym: EVEN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southern California Desert Retina Consultants, MC (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVEN Study
Record Dates: First submitted 2012-11-02; First posted 2012-11-07 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Submacular Vascularized Pigment Epithelial Detachments
Keywords: PED; AMD; CNV
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept (Other): All subjects will receive aflibercept
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Aflibercept

SUMMARY:
This study will evaluate the use of intravitreal aflibercept (anti-VEGF therapy) in patients with a type of macular degeneration known as vascularized pigment epithelial detachment. Previous studies have shown a generally poor outcome in treating this difficult to treat form of wet macular degeneration. More recently, multiple pilot studies have shown positive benefits to using anti-VEGF therapy. This study will evaluate the safety and efficacy of treating vascularize pigment epithelial detachment associated with wet macular degeneration with intravitreal aflibercept injection.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 50 years of age
* Subject is willing to participate in this study and to follow the criteria and protocol of this study.
* The study eye is treatment naïve regarding treatment of neovascular AMD.
* Subject is not involved with another clinical study currently.
* Subject is willing to follow the protocol outlined in the study.
* Ability to understand the informed consent and willingness to sign the informed consent.
* Presence of a submacular vascularized or fibrovascular PED. The investigator must search for the characteristic features of a vascularized PED summarized here:

  1. A notch of irregularity associated with an orange-yellow round, oval, or bean-shaped elevation of the RPE with a smooth, convex surface is seen on examination and fundus photography (FP). Fluorescein angiography (FA) shows uniform staining of the PED with a well-defined margin, and more intense staining (hot-spot) for the focus of the CNV.
  2. A fibrovascular PED with occult neovascularization typically shows stippled hyperfluorescence in the early phase with increasing hyperfluorescent staining and leakage in later phases of FA and a variable surrounding margin. There may be RPE folds.
  3. Regarding PED with a component of retinal angiomatous proliferation (RAP), the early features on FP including intraretinal neovascularization (IRN) frequently with adjacent small retinal hemorrhages in its lateral expansion in an irregularly stellate pattern before the development of retinal-choroidal anastomosis and the eventual PED in the later phases. The investigator is required to perform indocyanine-green (ICG) angiography at baseline to establish a RAP lesion and to rule-out polypoidal vasculopathy lesions, since the FA images may not be distinct.
  4. The investigator must also search for other features associated with a PED indicating the presence of a vascular component, i.e. hemorrhage, exudates, and/or chorioretinal folds.
  5. The investigator must confirm the presence of a PED on FA/FP and OCT. Spectral Domain OCT will be utilized. Specifically, the Spectralis OCT manufactured by Heidleberg to maintain uniformity for all the sites. The PED height, SA, GLD, and volume will be measured from the OCT images. The characteristic OCT findings of the vascularized PED must be confirmed, including a distinct elevation of the highly hyperreflective RPE layer with mild backscattering of the underlying choroidal layer in the portion of the PED without any CNV. For the portion of the PED with underlying CNV, typical OCT findings consist of moderate hyperreflectivity contiguous to the overlying markedly hyperreflective detached RPE corresponding to the CNV that usually extends to the choroidal layer. Besides the OCT characteristics confirmation must be made on the FP/FA images of the vascularized PED, as outlined above in detail.
* Central foveal involvement by the PED or the CNV due to age-related macular degeneration (AMD). The CNV may be classic, occult, or mixed, as long as it is associated with a PED. The CNV may be within the PED or adjacent to the margin of the PED.
* PED ≤ 12 disc area in size.
* BCVA with ETDRS of ≥ 19 letters and ≤ 73 letters (20/400 to 20/40).
* Evidence of submacular fluid outside or surrounding the PED.
* Surface area of the submacular hemorrhage needs to be < 50% of the entire PED.
* Submacular fibrosis needs to be < 50% of the entire PED.
* Sufficiently clear media (cornea, anterior chamber, lens, vitreous) for OCT, FA and FP.
* Intraocular pressure (IOP) of 25mmHg or less in the study eye, with or without use of ocular hypotensive agents.
* Prior treatment of neovascular AMD or any other forms of neovascularization in the fellow eye, including anti-VEGF or other forms of therapy targeted specifically for the fellow eye does not exclude the fellow eye from enrollment in this study. Prior focal corticosteroid treatment is allowed, as long as there is a lack of involvement of the study eye. However prior (within 90 days of Day 0) or current systemic corticosteroid therapy (oral or intravenous corticosteroid treatment) is not permitted.

Exclusion Criteria:

* Any prior treatment of neovascular AMD in eye for proposed enrollment (non-naïve eye), including previous anti-vascular endothelial factor (anti-VEGF) therapy, photodynamic therapy (PDT), radiation therapy, corticosteroid treatment, surgical treatment for CNV, thermal laser treatment, and any other prior treatment for neovascular AMD.
* Known serious allergies to aflibercept, fluorescein dye, drugs for pupillary dilation, topical anesthetic, sterilizing solution (e.g. Betadine Solution).
* Contraindication to pupillary dilation in study eye.
* Any condition (including inability to read visual acuity charts, or language barrier) that may preclude subjects ability to comply with the study protocol and requirements.
* Presence of any advanced systemic condition or end-stage disease, advanced Alzheimer Syndrome, end-stage cancer, etc., which will likely prevent subject from completing study.
* Previous therapeutic radiation in the region of the study eye.
* Prior retinal pigment epithelial (RPE) tear in study eye.
* Prior ocular surgery (except YAG laser capsulotomy) for study within the past 90 days.
* Anticipated ocular surgery (except YAG laser capsulotomy) for the next 12 months
* Prior therapy for AMD (except minerals and vitamins), including laser.
* Prior vitrectomy
* Presence of any causes of CNV and PED other than due to AMD.
* Presence of any substantial ocular disease (other than the CNV and PED) that may compromise vision in the study eye and/or confound interpretation of the data; e.g. substantial cataracts, concomitant diabetic retinopathy affecting the macula, advanced glaucoma, optic neuritis, optic neuropathy, or atrophy, marked macular atrophy, ocular vascular occlusion, history of retinal detachment, uveitis, viral or other forms of chorioretinitis, etc.
* Presence of ocular disease other than AMD affecting study eye, i.e. presumed ocular histoplasmosis syndrome, android streaks, pathologic myopia (spherical equivalent of ≥ -8 diopters of myopia or axial length of ≥ 25mm), choroidal rupture, multifocal choroiditis, etc.
* Active ocular infection (i.e., bacterial, viral, parasitic, or fungal) in either eye at screening
* Serous PED without neovascularization and polypoidal choroidal vasculopathy (PCV) lesions are excluded.
* Prior or current systemic anti-VEGF
* Prior (within 90 days of Day 0) or current corticosteroid therapy (oral or intravenous corticosteroid treatments).
* Sexually active men* or women of child-bearing potential** who are unwilling to practice adequate contraception during the study (adequate contraception measures include, stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly) *Contraception is not required for men with documented vasectomy. ** Post-menopausal women must be amenorrheic for at least 12 months in order not to be considered of child-bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 12 months
  Mean change in BCVA (Best Corrected Visual Acuity) from baseline measured at 4 meters on an ETDRS (Early Treatment Diabetic Retinopathy Study) chart at 12 months
Anatomic | 12 months
  Detailed anatomic descriptions and grading of lesion components and multi-modal anatomical changes (i.e. FP/FA, ICG, and OCT [Optical Coherence Tomography] findings) in a standardized fashion in a reading center setting at baseline and subsequent follow-up visits.

SECONDARY OUTCOMES:
Proportion of eyes reaching BCVA greater than or equal to 20/200 | 12 months
Proportion of eyes gaining greater than or equal to 0, 5, and 15 letters on ETDRS chart. | 12 months
Proportion of eyes losing greater than 5 and 15 letters on ETDRS chart | 12 months
Mean reduction in central macular thickness from baseline (central 1mm subfield) as measured on an OCT. | 12 Months
Mean changes in choroidal neovascular lesion (CNV) size on fluorescein angiography (FA) and fundus photography (FP) from baseline. | 12 months
Absence or complete resolution of subretinal fluid and cystoid macular edema. | 12 monts
Mean number of injections | 12 months
Status of fluorescein staining or leakage (increased or decreased) from baseline. | 12 months
Ocular safety outcome including ocular complications, i.e. RPE tears, uveitis, endophthalmitis | 12 months
Systemic safety outcome including cardiovascular events, cerebral vascular events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clement K Chan, M.D., Principal Investigator — Southern California Desert Retina Consultants
Locations (3):
- United States (3):
  - Jules Stein Eye Institute, Los Angeles, California
  - Southern California Desert Retina Consultants, Palm Desert, California
  - Black Hills Regional Eye Institute, Rapid City, South Dakota